CLINICAL TRIAL: NCT00010257
Title: Phase II Study Of Carboplatin Plus Paclitaxel Treatment Of Advanced Thymoma Or Thymic Carcinoma
Brief Title: Carboplatin Combined With Paclitaxel in Treating Patients With Advanced Thymoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000068461; U10CA021115 (NIH); E1C99 (Other: Eastern Cooperative Oncology Group (ECOG))
Record Dates: First submitted 2001-02-02; First posted 2003-01-27 (Estimated); Results first posted 2012-10-18 (Estimated); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Thymoma; Thymic Carcinoma
Keywords: thymoma; thymic carcinoma
MeSH Terms: conditions — Thymoma | interventions — Carboplatin; Paclitaxel; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Paclitaxel plus Carboplatin (Experimental): Paclitaxel 225 mg/m2 IV over 3 hours and Carboplatin AUC 6.0 IV over 30 minutes on day 1 of a 21-day cycle
  Interventions: Drug: carboplatin; Drug: paclitaxel

INTERVENTIONS:
Drug: carboplatin — Dosed to AUC of 6.0, given IV over 30 minutes day 1 of a 21-day cycle, for up to 6 cycles
  Other Names: CBDCA; Paraplatin; JM-8; NSC # 241240
Drug: paclitaxel — 225 mg/m2 given by intravenous (IV) infusion over 3 hours on day 1 of a 21-day cycle, for up to 6 cycles
  Other Names: Taxol; NSC #125973

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one chemotherapy drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of carboplatin combined with paclitaxel in treating patients who have advanced thymoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the objective response rate in patients with advanced thymoma or thymic carcinoma treated with carboplatin and paclitaxel.
* Determine the duration of response in these patients treated with this regimen.
* Determine the toxicity of this regimen in these patients.

OUTLINE: Patients receive paclitaxel by intravenous (IV) infusion over 3 hours followed by carboplatin IV over 30 minutes on day 1. Treatment repeats every 21 days for 2 courses in the absence of disease progression. Patients achieving complete or partial remission or stable disease receive 4 additional courses of therapy for a maximum of 6 courses. Further treatment may be given at the discretion of the treating physician.

Patients were followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 35-68 patients were to be accrued for this study within 3.8-4.6 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed invasive, recurrent, or metastatic thymoma or thymic carcinoma not amenable to potentially curative therapy by surgery
* Extensive disease (distant disease, pleural disease, pulmonary with or without mediastinal disease, or recurrent progressive disease in site of prior radiotherapy)
* Advanced limited disease allowed if ineligible for primary radiotherapy or surgery
* Measurable disease
* Age 18 and over
* ECOG Performance Status 0-1
* Granulocyte count at least 1,500 cells/mm^3
* Platelet count at least 100,000 cells/mm^3
* Bilirubin no greater than 1.5 mg/dL
* Creatinine no greater than 2.0 mg/dL
* Concurrent corticosteroids for myasthenia gravis or other chronic conditions allowed

Exclusion Criteria:

* Acute concurrent complications such as infection or post-surgical complications
* Other prior malignancy within the past 5 years unless curatively treated with no evidence of recurrence
* Pregnant or nursing. A negative pregnancy test was required, and fertile patients must use effective contraception
* Prior chemotherapy for metastatic disease. Prior preoperative or adjuvant chemotherapy allowed if disease-free survival prior to recurrence was more than 1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2001-06-19 (Actual); Primary Completion 2008-11 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick J. Loehrer, MD, Study Chair — Indiana University Melvin and Bren Simon Cancer Center
Locations (67):
- United States (67):
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - Joliet Oncology-Hematology Associates, Limited - West, Joliet, Illinois
  - Swedish-American Regional Cancer Center, Rockford, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Green Bay Oncology, Limited - Escanaba, Escanaba, Michigan
  - Dickinson County Healthcare System, Iron Mountain, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Meeker County Memorial Hospital, Litchfield, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology Hematology, PA - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - HealthEast Cancer Care at St. Joseph's Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - HealthEast Cancer Care at Woodwinds Health Campus, Woodbury, Minnesota
  - Minnesota Oncology Hematology, PA - Woodbury, Woodbury, Minnesota
  - Hunterdon Regional Cancer Center at Hunterdon Medical Center, Flemington, New Jersey
  - CCOP - Northern New Jersey, Hackensack, New Jersey
  - Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Aultman Cancer Center at Aultman Hospital, Canton, Ohio
  - Case Comprehensive Cancer Center, Cleveland, Ohio
  - MetroHealth Cancer Care Center at MetroHealth Medical Center, Cleveland, Ohio
  - St. Rita's Medical Center, Lima, Ohio
  - Mercy Fitzgerald Hospital, Darby, Pennsylvania
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Riddle Memorial Hospital Cancer Center, Media, Pennsylvania
  - Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania
  - Albert Einstein Cancer Center, Philadelphia, Pennsylvania
  - Hematology and Oncology Associates of Northeastern Pennsylvania, Scranton, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - Associates in Hematology-Oncology, PC at Crozer Regional Cancer Center, Upland, Pennsylvania
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - Green Bay Oncology, Limited at St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Gundersen Lutheran Cancer Center at Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
  - Froedtert Hospital and Medical College of Wisconsin, Milwaukee, Wisconsin
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin
  - Green Bay Oncology, Limited - Oconto Falls, Oconto Falls, Wisconsin
  - Marshfield Clinic - Indianhead Center, Rice Lake, Wisconsin
  - Green Bay Oncology, Limited - Sturgeon Bay, Sturgeon Bay, Wisconsin

REFERENCES:
- [Background] Loehrer PJ, Wang W, Aisner S, et al.: Long-term follow-up of patients with locally advanced or metastatic thymic malignancies: the Eastern Cooperative Oncology Group (ECOG) experience. [Abstract] J Clin Oncol 22 (Suppl 14): A-7050, 629s, 2004.
- [Result] Lemma GL, Lee JW, Aisner SC, Langer CJ, Tester WJ, Johnson DH, Loehrer PJ Sr. Phase II study of carboplatin and paclitaxel in advanced thymoma and thymic carcinoma. J Clin Oncol. 2011 May 20;29(15):2060-5. doi: 10.1200/JCO.2010.32.9607. Epub 2011 Apr 18. PMID 21502559

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was activated on February 21, 2001 and accrued its first patient on June 19, 2001. The thymoma stratum closed to accrual on March 27, 2007. The thymic carcinoma stratum closed to accrual on January 18, 2008.
Groups:
- Thymoma: Patients with diagnosis of thymoma
- Thymic Carcinoma: Patients with diagnosis of thymic carcinoma
Period: Overall Study
Arm/Group | Thymoma | Thymic Carcinoma
Started | 25 | 21
Completed | 24 | 21
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Thymoma | Thymic Carcinoma | Total
Number analyzed (Participants) | 25 | 21 | 46
Age, Continuous [Median (Full Range); unit: Years] | 50.8 [32.7 to 76.7] | 49.2 [20.8 to 67.1] | 50.7 [20.8 to 76.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 6 | 17
  Male | 14 | 15 | 29
Region of Enrollment [Number; unit: participants]
  United States | 25 | 21 | 46

OUTCOME MEASURES:

1. Primary Outcome: Best Overall Response by RECIST Criteria (Version 1.0)
Description: Number of eligible, treated participants in each response category by RECIST criteria
Time Frame: Assessed every 2 cycles (6 weeks)
Population: Analysis population included all eligible participants who received at least 1 dose of the protocol treatment
Measure: Number; unit: Participants
Arm/Group | Thymoma | Thymic Carcinoma
Number analyzed (Participants) | 23 | 20
Participants
  Complete Response | 3 | 0
  Partial Response | 5 | 6
  Stable Disease | 13 | 8
  Progression | 0 | 4
  Unevaluable | 2 | 2

2. Secondary Outcome: Duration of Response
Description: Time from first satisfaction of response criteria to onset of disease progression, assessed using RECIST criteria
Time Frame: assessed every 3 months for 2 years, then every 6 months for 3 years, then annually thereafter
Population: Number of participants achieving a complete or partial response by RECIST criteria
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Thymoma | Thymic Carcinoma
Number analyzed (Participants) | 8 | 6
Months | 16.9 [14 to NA] — The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment. | 5.0 [3.1 to 9.9]

ADVERSE EVENTS:
Time Frame: Assessed every 21 days while on treatment and for 30 days after the end of treatment.
Arm/Group | Thymoma | Thymic Carcinoma
Serious Adverse Events (participants affected / at risk) | 13/24 | 14/21
Other Adverse Events (participants affected / at risk) | 24/24 | 21/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Thymoma (N=24) | Thymic Carcinoma (N=21)
Anemia (Blood and lymphatic system disorders) | 1 | 2
Leukopenia (Blood and lymphatic system disorders) | 3 | 5
Neutropenia (Blood and lymphatic system disorders) | 8 | 6
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 2
Allergic Reaction (Immune system disorders) | 0 | 1
Cardiac, Other (Cardiac disorders) | 1 | 0
Fatigue (General disorders) | 2 | 6
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1
Blood Bilirubin Increased (Investigations) | 0 | 2
Febrile Neutropenia (Infections and infestations) | 0 | 2
Infection with grade 3-4 neutropenia (Infections and infestations) | 1 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0
Neuropathy - Sensory (Nervous system disorders) | 4 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Seizure (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Thymoma (N=24) | Thymic Carcinoma (N=21)
Anemia (Blood and lymphatic system disorders) | 17 | 19
Allergic Reaction (Immune system disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 13 | 12
Neutropenia (Blood and lymphatic system disorders) | 15 | 10
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 9
Edema (General disorders) | 2 | 2
Hypotension (Vascular disorders) | 2 | 0
Fatigue (General disorders) | 19 | 16
Fever (General disorders) | 2 | 3
Rigors/Chills (General disorders) | 0 | 2
Sweating (Skin and subcutaneous tissue disorders) | 1 | 2
Weight Gain (Metabolism and nutrition disorders) | 1 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 22 | 17
Nail Changes (Skin and subcutaneous tissue disorders) | 2 | 0
Pigmentation (Skin and subcutaneous tissue disorders) | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 3
Rash/Desquamation (Skin and subcutaneous tissue disorders) | 6 | 4
Anorexia (Metabolism and nutrition disorders) | 8 | 9
Constipation (Gastrointestinal disorders) | 3 | 3
Dehydration (Metabolism and nutrition disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 13 | 17
Stomatitis (Gastrointestinal disorders) | 3 | 7
Taste Disturbance (Gastrointestinal disorders) | 3 | 2
Vomiting (Gastrointestinal disorders) | 9 | 12
Diarrhea w/o Prior Colostomy (Gastrointestinal disorders) | 5 | 11
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Alkaline Phosphatase Increased (Investigations) | 1 | 7
Bilirubin Increased (Investigations) | 0 | 2
AST Increased (Investigations) | 5 | 6
ALT Increased (Investigations) | 4 | 5
Ataxia (Nervous system disorders) | 2 | 1
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 0 | 2
Dizziness/Lightheadedness (Nervous system disorders) | 3 | 2
Insomnia (Psychiatric disorders) | 4 | 3
Memory Loss (Nervous system disorders) | 0 | 2
Anxiety/Agitation (Psychiatric disorders) | 0 | 3
Neuropathy - Motor (Nervous system disorders) | 3 | 6
Neuropathy - Sensory (Nervous system disorders) | 23 | 16
Abdominal Pain (Gastrointestinal disorders) | 1 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 15 | 8
Chest Pain (Cardiac disorders) | 0 | 2
Headache (Nervous system disorders) | 3 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 14 | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 | 6
Creatinine Increased (Investigations) | 2 | 3
Urinary Frequency/Urgency (Renal and urinary disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No